CLINICAL TRIAL: NCT06925334
Title: Clinical Study Comparing Time to Glucose Attainment in Patients With Type 2 Diabetes Mellitus Treated With Degu Insulin Liraglutide Injection Versus Premixed Insulin
Brief Title: A Study Comparing Degu Insulin Liraglutide Injection With Premixed Insulin on the Prognosis of Diabetes Mellitus
Acronym: TLI vs PMI
Status: Enrolling by invitation | Phase: Phase 4 | Type: Interventional
Sponsor: Beijing Tsinghua Chang Gung Hospital (Other)
Collaborators: Taizhou First People's Hospital (Other); Wenzhou Central Hospital (Other); Wenzhou People's Hospital (Other); Chaohu Hospital of Anhui Medical University (Other); Affiliated Zhoushan Hospital of Wenzhou Medical University (Other); Yiwu Central Hospital (Other); Jinhua Municipal Central Hospital (Other); Dongyang People's Hospital (Other); The Central Hospital of Lishui City (Other); Affiliated Hospital of Jiaxing University (Other); Jinhua People's Hospital (Other); Wuhu City Second People's Hospital (Other); Affiliated Hospital of Nantong University (Other)
Responsible Party: Principal Investigator, ZHAO WENHUI, clinical professor, Beijing Tsinghua Chang Gung Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4.0 20240522
Record Dates: First submitted 2025-02-06; First posted 2025-04-13 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-02

CONDITIONS: Type 2 Diabetic Patients
Keywords: Tegu insulin liraglutide injection; Premixed human insulin or insulin analogues; Chinese patients with type 2 diabetes; time in range，TIR; Randomized Controlled Trial，RCT
MeSH Terms: interventions — insulin degludec

STUDY DESIGN:
Intervention Model Description: Randomized open, positive drug parallel control clinical study design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Treated with Degludec insulin (Experimental): Experimental group: Delgol insulin liraglutide injection
  Interventions: Drug: Degludec insulin
- Control group (No Intervention): Maintenance of original medication

INTERVENTIONS:
Drug: Degludec insulin — The pre-mixed human insulin or insulin analogues were stopped, and the treatment was switched to Delgol insulin liraglutide injection. The initial dose was subcutaneous injection of 80% (not more than 16 units) of the full daily dose of medium-acting insulin in the original insulin, once a day, and the dose of Delgol insulin liraglutide injection was adjusted according to the fasting blood glucose level. Example 1: If the patient is currently using Novorin 30 20iu bid, the conversion calculation is 40*70%*80%=22.4 units, which should be 16 units; In example 2, the patient applied eubrine 50 20 IU bid, and the conversion calculation was 40*50%*80%=16 units.
  Arms: Treated with Degludec insulin

SUMMARY:
A randomized open, positive parallel controlled clinical study design was adopted. Participants were randomly assigned 1:1 according to inclusion criteria and exclusion criteria into two treatment regiments: Delu insulin liraglupeptide injection group and premixed insulin (or premixed insulin analogue). After fasting blood glucose was controlled at 7.5mmol /l in the morning, blood glucose was monitored by CGM (14d), and the Time in Range (3.9-10 mmol/l) was compared. Glycated albumin was measured and stool samples were taken before treatment and at 4 weeks.

DETAILED DESCRIPTION:
Subjects eligible for inclusion press 1: 1. The proportion was randomly divided into the experimental group (Delu insulin liraglutide) and the control group (maintaining the original therapeutic drug). The first 14 days of the study was the dose adjustment period. The researchers timely adjusted the dosage of insulin or Delu insulin liraglutide according to the blood glucose monitoring results of the subjects, and the target value of blood glucose monitoring was set as fasting blood glucose <7.5 mmol/l in the morning. The average fasting blood glucose of the last 3 days of the previous 14 days is less than 7.5mmol/l to enter the next stage (if the blood glucose is not up to standard, the dose adjustment period can be extended for up to 7 days). After 14 days, the dose was stable. The blood glucose was monitored by CGM (14 days), and the Time in Range (3.9-10 mmol/l) was compared.

Experimental group: The pre-mixed human insulin or insulin analogues were stopped, and the treatment was switched to Delgol insulin liraglutide injection. The initial dose was subcutaneous injection of 80% (not more than 16 units) of the full daily dose of medium-acting insulin in the original insulin, once a day, and the dose of Delgol insulin liraglutide injection was adjusted according to the fasting blood glucose level. Example 1: If the patient is currently using Novorin 30 20iu bid, the conversion calculation is 40*70%*80%=22.4 units, which should be 16 units; In example 2, the patient applied eubrine 50 20 IU bid, and the conversion calculation was 40*50%*80%=16 units.

Control group: The original therapy was maintained until the 4th week.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily sign the informed consent form;
2. Male and female between the ages of 18 and 75 (inclusive);
3. Diagnosed with type 2 diabetes mellitus according to WHO standards (1999) for more than 6 months;
4. Those who use premixed human insulin or insulin analogues with or without oral hypoglycemic drugs (which cannot contain secretagogues and DPP4 inhibitors) >=3 months, and have poor blood sugar control;
5. Glycosylated hemoglobin > 7.0% and <=8.0% at screening;
6. Body mass index (BMI) > 18 kg/m^2 and <=35 kg/m^2;
7. Those who are willing and able to use the blood glucose meter for self-blood glucose monitoring according to the requirements of the program.

Exclusion Criteria:

1. People who are known to be allergic to Degu insulin or ingredients in its preparations;
2. Human glucagon-like peptide-1 (GLP-1) receptor agonist has been used within 3 months before screening;
3. Patients with hypoglycemic coma within 3 months before screening;
4. Patients with severe ketosis or ketoacidosis within 1 month before screening;
5. Severe complications of diabetes at the time of screening: such as severe proliferative diabetic retinopathy, a history of kidney transplantation, active peripheral vascular disease (such as diseases that have led to amputation, chronic foot ulcers, intermittent claudication, or require interventional procedures such as bypass or angioplasty);
6. Severe hypertension that cannot be controlled by treatment (defined as systolic blood pressure of not less than 180mmHg and/or diastolic blood pressure of not less than 100mmHg);
7. Patients with acute myocardial infarction, uncontrolled angina pectoris, uncontrolled arrhythmia, or severe heart failure (NYHA grading ≥III) in the 12 months prior to screening; New cerebrovascular accidents (including ischemic stroke, hemorrhagic stroke and transient ischemic attack) within 6 months prior to screening;
8. Liver and kidney function impairment: ALT, AST greater than 2.5 times the upper limit of normal, serum creatinine greater than 1.5 times the upper limit of normal;
9. Any conditions or co-existing diseases that the investigator determines may interfere with the test results, such as cardiovascular, respiratory, gastrointestinal, pancreatic, liver, kidney, nervous system, psychiatric, hematological (such as hematological tumors, hemolytic anemia, sickle cell disease, etc.), immune system, or other malignant tumors;
10. Mental disorder, unwilling to communicate or language barriers, unable to fully understand, cooperate and use the blood glucose meter;
11. Drugs that may have a significant effect on glucose metabolism, such as systemic corticosteroids, monoamine oxidase inhibitors, etc. are expected to be used within 3 months prior to screening;
12. Participated in other drug or device clinical studies 3 months before participating in this study;
13. Have a history of drug abuse and alcohol dependence in the past 5 years;
14. Known pregnancies (determined by pregnancy tests at the time of screening), women who are preparing to become pregnant or are lactating at the time of the test, or women of childbearing age who are unable to take adequate contraception (adequate contraception means Iuds, oral contraceptives and barrier measures);
15. Patients deemed unsuitable for participation in this study by the investigator;
16. Antibiotics and probiotics were used within 3 months before screening;
17. Family history of medullary thyroid cancer or medullary thyroid cancer or family history of MEN.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2024-05-20 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Time to blood glucose compliance | From the time of enrollment and signing of informed consent, the program started when blood glucose was controlled at 7.5 mmol/l for 14 days
  When morning fasting blood glucose was controlled at 7.5 mmol/l blood glucose was monitored using CGM to compare the time to reach blood glucose standard measured by CGM. Glucose attainment here is defined as a range of blood glucose control of 3.9-10 mmol/l

SECONDARY OUTCOMES:
GA（glycated albumin） | When subjects began 14 days of stable-dose insulin therapy, blood tests were performed at the end of treatment to measure glycated albumin
  High pressure liquid phase method was used for sample determination, and glycosylated albumin analyzer was used for sample determination according to SOP
Changes in intestinal flora | From enrollment until the end of the study, expected to be 28 days
  Changes in microflora were analyzed by 16SrRNA gene sequencing through the collection of stool samples at baseline and twice at the end of the dose stabilization period

CONTACTS AND LOCATIONS:
Overall Officials: WenHui ZHAO, Study Chair — Beijing Tsinghua Chang Gung Hospital
Locations (1):
- continuous glucose monitoring system（CGMS）, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No